CLINICAL TRIAL: NCT00000416
Title: Prevention of Arthritis-Related Work Disability: A Trial of Job Retention Services Provided to Employed Persons With Arthritis
Brief Title: Prevention of Arthritis-Related Work Disability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Boston University (Other)
Responsible Party: Principal Investigator, Saralynn J. Allaire, Professor, Boston University
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: P60AR020613 (NIH); P60AR020613 (NIH); NIAMS-012 (Other: Boston University); EEHRS Project 3 (Other: Boston University)
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Rheumatoid Arthritis; Systemic Lupus Erythematosus; Osteoarthritis, Knee; Ankylosing Spondylitis
Keywords: Arthritis; Rheumatic disorders; Work-related disability; Vocational rehabilitation (VR); Job retention services; Work limitations; Work instability
MeSH Terms: conditions — Arthritis, Rheumatoid; Lupus Erythematosus, Systemic; Osteoarthritis, Knee; Spondylitis, Ankylosing; Arthritis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rehabilitation counseling (Experimental): Rehabilitation counseling
  Experimental
  Rehabilitation counseling was provided by rehabilitation counselors. They administered the Work Experience Survey; provided and discussed disability rights and responsibilities and provided career counseling they as needed.
  Interventions: Other: Rehabilitation counseling
- printed information (Active Comparator): Active comparator
  Control group participants received relevant printed information in the mail only; no rehabilitation counseling
  Interventions: Other: Rehabilitation counseling

INTERVENTIONS:
Other: Rehabilitation counseling — Provided in 2 in-person meetings and in follow-up phone calls

SUMMARY:
People with rheumatic disorders (arthritis) often have trouble keeping their jobs. This study will look at whether vocational rehabilitation (VR) will improve the ability of employed people with arthritis to keep their jobs. Job retention VR services target key factors that increase the risk of job loss. They aim to modify jobs to reduce barriers caused by functional limitations and disease symptoms, future career planning, and establish a partnership with a VR counselor for ongoing help.

We will conduct the study among patients with rheumatic disorders recruited in eastern Massachusetts. We will give 120 study participants job retention services provided by VR counselors. We will give another 120 participants literature about employment- related resources. We will compare the outcomes of the two groups to evaluate the usefulness of job retention services in preventing job loss in people with rheumatic disorders.

DETAILED DESCRIPTION:
Job loss commonly occurs among people with rheumatic disorders. This study will determine whether vocational rehabilitation (VR) provided to employed people with rheumatic disorders will improve their ability to remain employed. VR is applied primarily to people who have already lost their jobs. However, using job retention VR services may prevent, or delay, the onset of employment work loss among people with rheumatic disorders. Job retention VR services target important employment-loss risk factors. They do so by modifying jobs to reduce barriers posed by functional limitations and symptoms, promoting future career planning, and establishing an alliance with a VR counselor for ongoing assistance.

The study is a randomized, controlled trial conducted among patients with rheumatic disorders recruited from the practices of rheumatologists in eastern Massachusetts.

We will randomly assign 120 study participants to receive job-retention services provided by VR counselors and 120 participants (controls) to receive literature about employment-related resources. We will assess intermediate outcome variables (self-efficacy, work limitations, and job accommodation-seeking behaviors) and the endpoint outcome variable, work instability (a measure that includes employment loss), immediately prior to the interventions and at 6-month intervals over a 24-month period after the interventions are carried out. We will compare the outcomes of the two groups to evaluate the usefulness of job retention services in forestalling work instability in this population.

ELIGIBILITY:
Inclusion Criteria:

* Must currently be employed full or part time
* Must live in selected communities in eastern Massachusetts

Exclusion Criteria:

* Plans to move from area
* Plans to have joint replacement surgery in next 6 months
* Plans to retire or go on disability within next 2 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 1997-09; Primary Completion 2001-08 (Actual); Study Completion 2001-08 (Actual)

PRIMARY OUTCOMES:
job losses | every 6 months for up to 42 months
  Periods of work cessation of at least 6 months.

SECONDARY OUTCOMES:
limitation in ability to work | every 6 months for up to 42 months
  Extent of on the job limitation due to health condition as measured by the Work Limitations Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Saralynn J. Allaire, Sc.D., Principal Investigator — Boston University
Locations (1):
- Boston University School of Medicine, Boston, Massachusetts, United States

REFERENCES:
- [Background] Allaire SH, Li W, LaValley,M: Work Problems reported by employed persons with reheumatic diseases and their association with work satisfaction. Arthritis Rheumatic 43:S128,2000
- [Background] Allaire SH, Li W, LaValley, M. Can job retention vocational rehabilitation services reduce work disability among employed persons with rheumatic diseases? Arthritis Rheum 44 (supplement):S813, 2001.
- [Background] Allaire SH. Update on work disability in rheumatic diseases. Curr Opin Rheumatol. 2001 Mar;13(2):93-8. doi: 10.1097/00002281-200103000-00001. PMID 11224732
- [Background] de Buck PD, Schoones JW, Allaire SH, Vliet Vlieland TP. Vocational rehabilitation in patients with chronic rheumatic diseases: a systematic literature review. Semin Arthritis Rheum. 2002 Dec;32(3):196-203. doi: 10.1053/sarh.2002.34609. PMID 12528084
- [Result] Allaire SH, Li W, LaValley MP. Reduction of job loss in persons with rheumatic diseases receiving vocational rehabilitation: a randomized controlled trial. Arthritis Rheum. 2003 Nov;48(11):3212-8. doi: 10.1002/art.11256. PMID 14613285
- [Result] Allaire SH, Niu J, Lavalley MP. Employment and Satisfaction Outcomes From a Job Retention Intervention Delivered to Persons with Chronic Diseases. Rehabilitation Counseling Bulletin 48(2):100-109, 2005